CLINICAL TRIAL: NCT06738368
Title: Dose-Adjusted Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin (DA-EPOCH) ± Rituximab + Recombinant Erwinia Asparaginase (JZP458; Rylaze®) for the Treatment of Newly-Diagnosed Adults With Philadelphia Chromosome-Negative Acute Lymphoblastic Lymphoma/Leukemia
Brief Title: Etoposide, Prednisone, Vincristine, Cyclophosphamide, and Doxorubicin (DA-EPOCH) With or Without Rituximab Plus Recombinant Erwinia Asparaginase (JZP458) for the Treatment of Newly Diagnosed Ph Negative B-Acute Lymphoblastic Leukemia or T Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124788; NCI-2024-09417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020869 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative; T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; Cyclophosphamide; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DA-EPOCH, rituximab, JZP458) (Experimental): Patients receive etoposide IV, doxorubicin IV and vincristine IV over 96 hours on days 1-4, cyclophosphamide IV over 1 hour on day 5, prednisone PO BID on days 1-5 of each cycle. In addition, CD20 positive patients receive rituximab IV on day 1 or 5 of each cycle. Patients also receive JZP458 IM every 2-3 days on days 7-21 for up to 7 doses. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 6, 7, or 8, patients also receive pegfilgrastim SC once or filgrastim SC QD until ANC > 2000/uL past nadir. Patients also undergo blood sample collection and bone marrow collection throughout the study. Additionally, patients with extramedullary disease may undergo CT or PET/CT throughout the study.
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Biological: Filgrastim; Biological: Pegfilgrastim; Procedure: Positron Emission Tomography; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given IM
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Collection — Undergo bone marrow sample collection
  Other Names: Collection, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given CIV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given CIV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine — Given CIV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial tests how well etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin (DA-EPOCH) with or without rituximab plus recombinant Erwinia asparaginase (JZP458) works in treating patients with newly diagnosed Philadelphia chromosome (Ph) negative B-acute lymphoblastic leukemia (ALL) or T-ALL. Chemotherapy drugs, such as etoposide, vincristine, cyclophosphamide and doxorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs, such as prednisone, lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. JZP458 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving DA-EPOCH with or without rituximab plus JZP458 may kill more cancer cells in patients with newly diagnosed Ph negative B-ALL or T-ALL.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive etoposide intravenously (IV), doxorubicin IV and vincristine IV over 96 hours on days 1-4, cyclophosphamide IV over 1 hour on day 5, prednisone orally (PO) twice daily (BID) on days 1-5 of each cycle. In addition, CD20 positive patients receive rituximab IV on day 1 or 5 of each cycle. Patients also receive JZP458 intramuscularly (IM) once every 2-3 days on days 7-21 for up to 7 doses. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Starting on day 6, 7, or 8, patients also receive pegfilgrastim subcutaneously (SC) once or filgrastim SC once daily (QD) until absolute neutrophil count (ANC) > 2000/uL past nadir. Patients also undergo blood sample collection and bone marrow collection throughout the study. Additionally, patients with extramedullary disease may undergo computed tomography (CT) or positron emission tomography (PET)/CT throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older) with newly-diagnosed Ph- B-ALL or T-ALL
* In the opinion of the treating investigator, patients must be an unsuitable candidate for a pediatric-inspired regimen, reasons for which may include (but not be limited to) older age (e.g., ≥ 40 years), practical/logistical barriers to or toxicity concerns from administration of a pediatric-inspired regimen
* Marrow or blood involvement by ALL detectable by multi-parameter flow cytometry (MFC)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. (Performance status of 3 will be allowed if poor performance status is thought to be directly secondary to ALL.)
* Total bilirubin ≤ 2.0 x upper limit of normal (ULN) (unless attributed to Gilbert's disease or other causes of inherited indirect hyperbilirubinemia, at which point total bilirubin must be ≤ 4.0 x ULN) (Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the total bilirubin is ≤ 5.0 x ULN and alanine aminotransferase [ALT]/aspartate aminotransferase [AST] are ≤ 8.0 x ULN.)
* AST (serum glutamic oxaloacetic transaminase [SGOT])/ALT (serum glutamic pyruvic transaminase [SGPT]) ≤ 5.0 x institutional ULN. (Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the total bilirubin is ≤ 5.0 x ULN and ALT/AST are ≤ 8.0 x ULN.)
* Calculated creatinine clearance of ≥ 60 ml/min/1.73 m^2, as measured by the Modification of Diet in Renal Disease (MDRD) equation, will be eligible
* As patients with ALL frequently have cytopenias, no hematologic parameters will be required for enrollment or to receive the first cycle of treatment. However, adequate recovery of blood counts will be required to receive subsequent cycles
* Ability to give informed consent and comply with the protocol
* Anticipated survival of at least 3 months, independent of ALL
* Female subjects of childbearing potential should use effective non-hormonal contraceptive methods during treatment with JZP458 and for 3 months after the last dose of study drug. Male subjects with female partners of childbearing potential must agree to use an effective method of birth control from the time of signing the consent form until at least 3 months after the last dose of study drug

Exclusion Criteria:

* Prior systemic therapy for ALL except to control acute symptoms and/or leukocytosis (e.g., corticosteroids, cytarabine, etc.). Cytarabine 500 mg/m^2 per dose up to 2 doses and/or the equivalent of prednisone 50 mg/m^2/day for up to 2 days are permitted
* Burkitt lymphoma/leukemia
* Isolated extramedullary or known parenchymal central nervous system (CNS) disease
* Known hypersensitivity or intolerance to any of the agents under investigation
* Known history of grade 3+ pancreatitis or chronic pancreatic insufficiency
* Known active chronic liver disease including, but not limited to, non-alcoholic steatohepatitis, cirrhosis, or non-alcoholic fatty liver disease
* Other medical or psychiatric conditions that in the opinion of the investigator would preclude safe participation in the protocol
* Pregnant or nursing

  * Pregnancy test is only required in women, unless they are highly unlikely to conceive (defined as [1] surgically sterilized, or [2] postmenopausal [i.e., a woman who is > 50 years old or who has not had menses for ≥ 1 year], or [3] not heterosexually active)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Measurable residual disease (MRD) negativity | After 4 cycles of treatment (cycle length = 21 days)
  Will be measured by multi-parameter flow cytometry (MFC). Will be assessed according to the National Comprehensive Cancer Network response criteria.

SECONDARY OUTCOMES:
MRD negativity | After 1 cycle of study therapy (cycle length = 21 days)
  Will be measured by MFC. Will be assessed descriptively, using means, medians, and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures.
Incidence of grade 3 or higher non-hematologic adverse events (AEs) | Up to 30 days after last dose of study treatment
  Will be assessed descriptively, using means, medians, and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures. The incidence of AEs will be reported as ratios or percentages.
Event-free survival (EFS) | Up to 5 years
  Will be assessed descriptively, using means, medians, and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures. Kaplan-Meier curves will be used to depict EFS.
Relapse-free survival (RFS) | Up to 5 years
  Will be assessed descriptively, using means, medians, and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures. Kaplan-Meier curves will be used to depict RFS.
Overall survival (OS) | Up to 5 years
  Will be assessed descriptively, using means, medians, and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures. Kaplan-Meier curves will be used to depict OS.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan D. Cassaday, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No